CLINICAL TRIAL: NCT02554942
Title: An Open-Label Study of the Safety Of NeoRecormon in Patients With Solid Tumors Being Treated With Platinum Capable of Inducing Anemia
Brief Title: A Study of Epoetin Beta (NeoRecormon) in Participants With Solid Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17912
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (1):
- Epoetin beta (Experimental): Participants will receive weekly SC injection of epoetin beta (450 international units per kilogram [IU/kg]) for 16 weeks.
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — Participants will receive weekly SC injections of epoetin beta beginning at 450 IU/kg, with doses adjusted according to hemoglobin level. Treatment will continue for a total of 16 weeks.
  Other Names: NeoRecormon

SUMMARY:
This study will evaluate the safety of subcutaneous (SC) epoetin beta (NeoRecormon) in adults with solid tumors being treated with platinum-based chemotherapy capable of inducing anemia. The anticipated time on study treatment is 16 weeks, and the target sample size is approximately 208 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Presence of solid tumor(s)
* Receiving platinum-based therapy capable of inducing anemia

Exclusion Criteria:

* Red blood cell transfusion within 7 days prior to study drug
* Relevant acute or chronic bleeding requiring therapy within 3 months prior to study drug
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 16 weeks

SECONDARY OUTCOMES:
Hemoglobin response rate index | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (10):
- Spain (10):
  - Alcoy
  - Barakaldo
  - Barcelona
  - Cáceres
  - El Palmar Murcia
  - Manresa
  - Salamanca
  - San Cristóbal de La Laguna
  - Valencia
  - Zaragoza